CLINICAL TRIAL: NCT04389112
Title: Study of Metabolic Changes in the Transformation Malignant Precancerous Skin Lesions
Acronym: MITOSKIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2019/3
Record Dates: First submitted 2020-03-31; First posted 2020-05-15 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Cutaneous Squamous Cell Carcinoma; Basal Cell Carcinomas
Keywords: Actinic keratosis; mitochondria; metabolism
MeSH Terms: conditions — Carcinoma, Basal Cell; Keratosis, Actinic | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients with actinic keratoses (Experimental)
  Interventions: Other: biopsy
- patients with squamous cell carcinoma in situ (Experimental)
  Interventions: Other: biopsy
- patients with squamous cell carcinomas (Experimental)
  Interventions: Other: biopsy
- patient with invasive metastates (Experimental)
  Interventions: Other: biopsy

INTERVENTIONS:
Other: biopsy — Skin biopsies will be performed according to standard practices in the usual aseptic conditions, the operator wearing sterile gloves. A circular knife 3 mm will be used. Procedure interventions do not involve a drug or a device.

SUMMARY:
Skin carcinomas are the most frequent cancers in the world, including basal cell carcinomas and cutaneous squamous cell carcinoma (cSCCs), with more than 60.000 new annual cases in France. Their incidence increases mainly due to ultraviolet (UV) exposure and population ageing. Then from 1994 to 2006, the incidence of cSCC has increased by 300%. CSCCs typically manifests as a spectrum from a precursor actinic keratosis (AK) - possible spontaneous regression at this stage- to in situ cSCC invasive cSCC and finally metastatic cSCC.

DETAILED DESCRIPTION:
Although growing evidence indicates that bioenergetic metabolism plays an important role in the progression of tumorigenesis, little information is available on the contribution of reprogramming of energy metabolism in cancer initiation and how it influences further the bioenergetic behavior of tumors.

By applying a quantitative proteomic approach, the consortium has recently found that specific metabolic modifications precede cSCC.

This study will investigate the role of energy metabolism in malignant transformation of premalignant skin lesions into cSCC, and in cSCC progression, with correlation with clinical characteristics and metastatic outcomes. Using several cutting-edge technologies in human samples, the team will evaluate whether targeting energy metabolism has the potential to be used as curative treatments for cSCC and whether pre-determined metabolic alterations could be exploited as new preventive strategies. These modifications in energy metabolism could be used as prognostic and diagnostic biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Every patient with suspected lesion :

  * AK,
  * in situ cSCC,
  * infiltrative cSSC
  * cSCC with recurrent disease
  * cSCC with cutaneous metastases.
* Patients 18 years of age or older,
* Patients with suspected AK or BCC lesions (in situ, infiltrating or metastatic),
* Patient able to sign a consent form,
* Patient affiliated with a Social Security system.

Exclusion Criteria:

* Prior systemic treatment such as checkpoint inhibitors or chemotherapy.
* Patients with cSCC or AK localized on visible zone of the face or folds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-02-28 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who have a glycolysis profile (proteomic analysis liquid chromatography-mass spectrometry (LC-MS/MS)) | Day 1
  Metabolic profiling of different stages of carcinogenesis: glycolysis, oxidative phosphorylation
Proportion of patients who have an oxidative profile (proteomic analysis liquid chromatography-mass spectrometry (LC-MS/MS)) | Day 1
  Metabolic profiling of different stages of carcinogenesis: glycolysis, oxidative phosphorylation

SECONDARY OUTCOMES:
Evaluation of skin differentiation markers | Day 1
  % of samples in each category (AK, in situ, ...) that present differentiation features are assessed by immunostaining of loricrin, filaggrin, K10
Evaluation of cSCC aggressiveness markers | Day 1
  % of samples expressing aggressive markers will be assessed by evaluating the proliferation index, degree of differentiation, invasion beyond subcutaneous fat, perineural invasion, vascular invasion level of infiltration following immunohistochemistry analyses on formalin-fixed paraffin-embedded tissue sections.
Evaluation of skin apoptotic markers | Day 1
  % of samples with high apoptotic cell death level will be assessed by immunostaining using antibody against cleaved caspase-3.
Evaluation of mitochondrial metabolism on skin biopsies | Day 1
  % of samples with high mitochondrial activity will be evaluated by comparing oxygen consumption rate by different fresh samples.
Evaluation of cancer proliferative features on skin biopsies | Day 1
  % of samples that are highly proliferative will be calculated by measuring the ability of colony formation (SRB Test) and cell cycle progression (flow cytometer, western).

CONTACTS AND LOCATIONS:
Overall Officials: Marie BEYLOT-BARRY, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Hôpital Saint-André - CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Obre E, Rossignol R. Emerging concepts in bioenergetics and cancer research: metabolic flexibility, coupling, symbiosis, switch, oxidative tumors, metabolic remodeling, signaling and bioenergetic therapy. Int J Biochem Cell Biol. 2015 Feb;59:167-81. doi: 10.1016/j.biocel.2014.12.008. Epub 2014 Dec 24. PMID 25542180
- [Background] Hosseini M, Dousset L, Mahfouf W, Serrano-Sanchez M, Redonnet-Vernhet I, Mesli S, Kasraian Z, Obre E, Bonneu M, Claverol S, Vlaski M, Ivanovic Z, Rachidi W, Douki T, Taieb A, Bouzier-Sore AK, Rossignol R, Rezvani HR. Energy Metabolism Rewiring Precedes UVB-Induced Primary Skin Tumor Formation. Cell Rep. 2018 Jun 19;23(12):3621-3634. doi: 10.1016/j.celrep.2018.05.060. PMID 29925003
- [Background] Hosseini M, Dousset L, Michon P, Mahfouf W, Muzotte E, Bergeron V, Bortolotto D, Rossignol R, Moisan F, Taieb A, Bouzier-Sore AK, Rezvani HR. UVB-induced DHODH upregulation, which is driven by STAT3, is a promising target for chemoprevention and combination therapy of photocarcinogenesis. Oncogenesis. 2019 Sep 24;8(10):52. doi: 10.1038/s41389-019-0161-z. PMID 31551419
- [Background] Mahfouf W, Hosseini M, Muzotte E, Serrano-Sanchez M, Dousset L, Moisan F, Rachidi W, Taieb A, Rudolf J, Rezvani HR. Loss of Epidermal HIF-1alpha Blocks UVB-Induced Tumorigenesis by Affecting DNA Repair Capacity and Oxidative Stress. J Invest Dermatol. 2019 Sep;139(9):2016-2028.e7. doi: 10.1016/j.jid.2019.01.035. Epub 2019 Mar 13. PMID 30878676